CLINICAL TRIAL: NCT06035419
Title: The Effect of Training Given to Immigrant Primiparous Mothers in the Neonatal Intensive Care Unit on Breastfeeding Success
Brief Title: The Effect of Breastfeeding Education to Immigrant Mothers in the NICU on Breastfeeding Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sibel Serap Ceylan, Associate professor, PhD, RN, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PAU SBF
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Breastfeeding; Immigrant
Keywords: Breast milk; Neonatal intensive care; Immigrant; Breastfeeding; Education
MeSH Terms: conditions — Breast Feeding | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: randomized-controlled and single-blind study
Who Masked: Participant
Masking Description: In order to avoid bias in the study, a nurse who was not involved in the study performed the LATCH scoring and evaluation of the suckling time and feeding style of the infants, without knowing which group the mothers were in. In addition, mothers to be included in the experimental and control groups were determined by simple randomization method in order to prevent selection bias in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education (Experimental): A specially prepared training program for immigrant mothers was applied to the mothers in the experimental group.
  Interventions: Other: education
- control (No Intervention): No interventions were made to the control group other than the routine interventions of the clinic (unstructured training practices given by the individual effort of the nurse).

INTERVENTIONS:
Other: education — breastfeeding education for migrant mothers
  Other Names: breastfeeding education
  Arms: education

SUMMARY:
Feeding the infant with breast milk in neonatal intensive care units is essential. However, breastfeeding can be adversely affected in this complex environment, especially for immigrant mothers. In order to ensure the success of breastfeeding in the neonatal intensive care unit, education and support of the mother are required. While doing this, structured and planned education programs should be implemented taking into account the individual characteristics of the mother (culture, age, etc.).This study aimed to evaluate the effect of education given to immigrant mothers on breastfeeding success of mothers. The study was a randomized controlled, single-blind clinical trial.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of education given to immigrant mothers on breastfeeding success of mothers.

Method: In this randomized-controlled, single-blind study, 80 immigrant mothers (40 intervention groups, 40 control groups) were recruited.

The study included primiparous immigrant mothers whose mother tongue was not Turkish, whose baby was hospitalized for the first time in the NICU, whose baby was born at 34-40 weeks of gestation, whose baby was fed orally, and whose suckling was not impaired.

In the study, 40 participants were included in the experimental group and 40 participants in the control group. At the end of the study, Cohen's d was calculated to determine the effect size and was found to be 1.80.

A simple randomization method was used to randomly assign the mothers included in the study to the experimental and control groups. To avoid bias in the study, a nurse who was not involved in the study made the LATCH scoring and evaluation of the suckling time and feeding style of the infants, without knowing which group the mothers were in. In addition, mothers to be included in the experimental and control groups were determined by a simple randomization method to prevent selection bias in the study.

Mother-baby information form, Nutrition follow-up form, and LATCH were used to collect the study data.

The mothers to be included in the study were informed by an interpreter before the study and their consent was obtained. It was ensured that the mothers in both groups answered the questions in the data collection forms through a translator. Information about the baby was taken from the patient's file.

A specially prepared training program for immigrant mothers was applied to the mothers in the experimental group. In the control group, no interventions were made except for the routine interventions of the clinic (unstructured training practices given by the individual effort of the nurse).

The first of the parameters used to evaluate breastfeeding success is the mothers' LATCH score averages. LATCH scores of mothers were evaluated by observation. LATCH evaluations of the mothers in the experimental group were made at the first breastfeeding before the training and on the 1st, 2nd, and 3rd days after the training. The LATCH evaluations of the control group were made at the first breastfeeding and on the 1st, 2nd, and 3rd days.

Another parameter examined to evaluate breastfeeding success is the suckling time of babies at each breastfeeding. The suckling time of the babies was measured with a stopwatch at each feeding.

The last of the parameters to evaluate breastfeeding success is the feeding style of infants. Information about the feeding style of infants was obtained from the nurse observation form.

ELIGIBILITY:
Inclusion Criteria:

* Immigrant mothers whose baby was hospitalized for the first time in the NICU, whose baby was born at 34-40 weeks of gestation, whose baby was fed orally and who did not prevent suckling, whose mother tongue was not Turkish, and who volunteered to participate in the study.

Exclusion Criteria:

* Migrant mothers whose babies were hospitalized in the NICU before, whose baby was younger than 34 weeks of gestation, whose baby was not fed orally, who were not primiparous, and who did not volunteer to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
LATCH score | 3 days
  LATCH was used to evaluate breastfeeding success. Each item is evaluated between 0-2 points. The total score that can be obtained from the vehicle is 10, and a high score means high breastfeeding success. Evaluation is done through observation.
sucking time of babies | 3 days
  To evaluate the suckling time of babies, sucking time was measured with a stopwatch at each feeding.
feeding type of babies | 3 days
  Information about the feeding style of infants was obtained from the nurse observation form. The characteristics for the type of nutrition are; breastfeeding only, spoon feeding only, spoon feeding and breastfeeding together.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)